CLINICAL TRIAL: NCT04087304
Title: Prospective Validation of a Hip and Knee Scoring System to Predict Complication Rate and Candidacy for Total Hip and Knee Arthroplasty
Brief Title: Hip and Knee Scoring System to Predict Complication Rate and Candidacy for Total Hip and Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started, no participants enrolled. Study was closed at Rush
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brett Levine, MD, Associate Professor, Rush University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 18081101-IRB01
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Risk Group (No Intervention)
- Mild Risk Group (No Intervention)
- Moderate Risk Group (Active Comparator)
  Interventions: Behavioral: Risk Status Optimization
- High Risk Group (Active Comparator)
  Interventions: Behavioral: Risk Status Optimization

INTERVENTIONS:
Behavioral: Risk Status Optimization — Assessment of risk factors putting surgical candidates of total hip and knee arthroplasty at higher risk of complication, and promoting risk factor optimization, thereby decreasing associated risk.
  Arms: High Risk Group; Moderate Risk Group

SUMMARY:
This study is a prospective validation study of a new hip and knee replacement-specific questionnaire that can be used to predict postoperative complications. The purpose of this study is to confirm the validity of a new hip and knee scoring system to be used as a clinical tool to predict potential complication rates in patients undergoing total hip or knee replacement surgery. This scoring system aims to stratify patients into specific risk categories based a standardized calculated score. Patients will be evaluated on health risk factors and severity of disease on radiographic imaging prior to surgery, associated to higher complication rates following surgery. The hopeful anticipated result of this study is a prospective validation of the scoring system with both statistical and clinical significance in predicting postoperative complication rates in patients with moderate to high health risk,

This stratification system may prove meaningful by allowing these patients, especially those classified as High-Risk, to be incorporated into more appropriate healthcare bundle payment systems that account for their higher financial demands. Furthermore, the stratification may allow for preoperative counseling and a shift towards non-operative management, or surgeon-patient conversations regarding the need to modify a portion of their objective risks prior to surgical intervention. Predictive risk models such as the one presented in the current study will be essential tools as the number of total hip arthroplasty procedures performed each year continue to increase and both the numbers of procedures and associated complications impose a significant cost on the U.S. healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be male or female of any race.
2. Patients much be age greater than 18 years old.
3. Patients undergoing a primary total hip arthroplasty (THA) or total knee arthroplasty (TKA) by participating surgeons at this institution.

Exclusion Criteria:

1. Patients with history of native joint infection or active periprosthetic infection according to Musculoskeletal Infection Society (MSIS) Criteria.
2. Patients requiring removal of hardware during their primary total hip arthroplasty (THA) or total knee arthroplasty (TKA).
3. Patients requiring use of revision THA or TKA components (stems, augments).
4. Patients with history of neuromuscular disorder impairing ability to participate in standard postoperative rehabilitation protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Optimized Risk Factors | Optimization time period covers a total time period of 6 months.
  A Scoring System Questionnaire with risk factors associated with increased risk of complications in patients undergoing total hip and knee arthroplasty will be collected
  Risk factors collected include obesity, drug allergies, presence of osteophytes, soft tissue to patella thickness, flexion contracture, diabetes, chronic opioid use, co-morbidities, prior knee surgeries, etiology of arthritis, smoking status, and reported disability. Each are measured on a scale of -5 to 10, with 10 being the best outcome. All the risk factors are added together and that comprises the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No